CLINICAL TRIAL: NCT03427788
Title: Randomized, Placebo-controlled, Double-blind, Parallel Group Study to Investigate the Safety, Tolerability and Pharmacokinetics of Increasing Single Oral Doses of BAY2328065 Including the Relative Bioavailability Between Solution and Tablet Formulation and the Effect of Food on the Pharmacokinetics of BAY2328065 in Healthy Men
Brief Title: BAY2328065 Single Dose Escalation, Safety and Tolerability, Pharmacokinetics, Relative Bioavailability, Food Effect
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 19250; 2017-004056-38 (EudraCT Number)
Record Dates: First submitted 2018-02-05; First posted 2018-02-09 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum (Experimental): Study group 1-11 of BAY2328065 (increasing dose levels for study group 2-11)
  Interventions: Drug: BAY2328065
- Placebo (Placebo Comparator): Study group 1-11 of Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BAY2328065 — Doses from 2.25-700 mg once daily in an escalating manner as liquid service formulation (LSF) or tablets
  Arms: Verum
Drug: Placebo — Matching placebo, once daily in an escalating manner as LSF or tablets
  Arms: Placebo

SUMMARY:
This single center, double-blind, randomized study with up to 11 treatment groups evaluates the safety and tolerability, pharmacokinetics, relative bioavailability and food effect of single ascending doses of BAY2328065

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers, aged 18 - 45 years
* Body mass index (BMI): 18 ≤ BMI ≤ 30 kg/m²
* Smoking less than 10 cigarettes / day
* Signed informed consent
* Use of an accepted method of contraception for the duration of the study.

Exclusion Criteria:

* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders, thyroid disorders or malignant tumors
* Known severe allergies, non allergic drug reactions, or multiple drug allergies
* Medication history: any regular medication, esp. drugs known to induce/inhibit liver enzymes or transporters
* Clinically relevant findings in physical examination; ECG, blood pressure; laboratory values

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2018-03-21 (Actual); Primary Completion 2018-10-29 (Actual); Study Completion 2019-02-11 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | Up to 8 days
  The frequency of adverse events collected from dosing until follow up, i.e. 8 days after dosing
Severity of treatment-emergent adverse events | Up to 8 days
  The severity of adverse events collected from dosing until follow up, i.e. 8 days after dosing
  Severity is assessed by the following criteria:
  1. Results in death
  2. Is life-threatening
  3. Requires inpatient hospitalization or prolongation of existing hospitalization
  4. Results in persistent or significant disability / incapacity
  5. Is a congenital anomaly / birth defect
  6. Is another serious or important medical event as judged by the investigator

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Berlin GmbH, Berlin, Germany